CLINICAL TRIAL: NCT03400371
Title: Biology of Juvenile Myoclonic Epilepsy
Acronym: BIOJUME
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); Charles University, Czech Republic (Other); Hopital Universitaire Robert-Debre (Other); Vestre Viken Hospital Trust (Other); The Hospital for Sick Children (Other); Cardiff University (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 199351; CIHR ID: MOP-142405 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2017-11-20; First posted 2018-01-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Juvenile Myoclonic Epilepsy
Keywords: JME; Epilepsy; Juvenile Myoclonic Epilepsy; Genomewide Association Study; Genetics
MeSH Terms: conditions — Myoclonic Epilepsy, Juvenile; Epilepsy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients diagnosed with JME: People who meet the eligibility requirements and have been diagnosed with juvenile myoclonic epilepsy.
  Interventions: Other: Blood draw
- Controls: People without a lifetime history of seizures.
  Interventions: Other: Existing samples

INTERVENTIONS:
Other: Blood draw — Participation includes one visit for one blood draw per recruited patient. 10-20ml peripheral venous blood will be taken from the antecubital fossa. The DNA from the blood sample will then be extracted and resequenced for analysis.
  Groups: Patients diagnosed with JME
Other: Existing samples — Control DNA samples will be used that have been previously acquired in other studies.
  Groups: Controls

SUMMARY:
The investigators are collecting genetic information through blood samples as well as clinical and EEG data from over 1000 people with Juvenile Myoclonic Epilepsy (JME) across the UK, Europe and North America. This study will draw on both existing and new samples from JME patients. These will be compared to anonymised data from samples for 2000 controls. The goal of this study is to find the genetic cause of JME. Finding the cause will help create better treatments for JME, as well as improve patient outcomes by allowing us to detect it earlier.

DETAILED DESCRIPTION:
Epilepsy is a common neurological disorder affecting 1% of the population. There are over 30 types of epilepsy, some common, some rare. Most epilepsies arise in childhood and have a genetic cause. Approximately 40% of patients have the common forms of Genetic Generalised Epilepsy (GGE), and the commonest GGE is "Juvenile Myoclonic Epilepsy" or JME.

The goal of this study is to find the genetic cause for JME. The investigators will do this by comparing the genetic code in JME patients with that in people who do not have epilepsy. This study will use clues from their electroencephalograph or brainwave test that is used to help diagnose epilepsy. Participants will provide a single blood sample, along with permission to collect clinical data about their diagnosis and a copy of their clinical EEG. There is no direct benefit or risk to the research participants but the results from this study may help other people with epilepsy or brain impairments in the future.

There is overwhelming evidence that JME is caused by changes in genetic code. These changes are likely to be found in more than just one gene and there may be more than one type of change. In order to find these changes, this study will look at a large number of people with JME and compare their genetic code with people who do not have epilepsy. Finding the causes of JME will lead to better understanding of its cause, new treatments, and tailoring of treatments according to a person's genetic make-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Juvenile Myoclonic Epilepsy in accordance with Consensus criteria

  * Age of myoclonus onset 10-25 years
  * Seizures comprising predominant or exclusive early morning myoclonus of upper extremities
  * EEG interictal generalized spikes and/or polyspike and waves with normal background
* Current age 10-40 years

Exclusion Criteria:

* Myoclonus only associated with carbamazepine or lamotrigine therapy
* EEG showing predominant focal interictal epileptiform discharges or abnormal background
* Any evidence of progressive or symptomatic myoclonus epilepsy or focal seizures
* Global learning disability
* Dysmorphic syndrome
* Unable to provide informed consent

Regrettably, we are currently unable to accept self-referrals to the BIOJUME study.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: People in the UK, Europe, and North America with a diagnosis of Juvenile Myoclonic Epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Genomewide DNA association study | Day 1
  Association between SNP marker and phenotype is measured using genomewide DNA markers, which enables us to test support for molecular networks that act on seizure susceptibility

SECONDARY OUTCOMES:
Quantitative EEG endophenotype | Day 1
  Brain network ictogenicity is measured using quantitative EEG data

CONTACTS AND LOCATIONS:
Overall Officials: K Pal, MD PhD, Principal Investigator — King's College London
Locations (15):
- United States (3):
  - Mount Sinai-Beth Israel Medical Center, New York, New York
  - St Luke's Roosevelt Hospital, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
- Hospital for Sick Kids, Toronto, Ontario, Canada
- Charles University, Prague, Czechia
- Danish National Epilepsy Centre, Dianalund, Denmark
- Tallinn Children's Hospital, Tallinn, Estonia
- University Robert Debré, Paris, France
- Commissione Genetica Lega Italiana contro l'Epilepssia, Roma, Italy
- Vestre Viken Health Trust, Oslo, Drammen, Norway
- United Kingdom (5):
  - Walton Centre for Neurology and Neurosurgery, Liverpool
  - Royal London Hospital, London
  - St Thomas' Hospital, London
  - King's College Hospital NHS Trust, London
  - Swansea University, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Childhood Epilepsy website — https://childhoodepilepsy.org